CLINICAL TRIAL: NCT02676635
Title: National Center for Construction Safety and Health Research and Translation: Safety Voice for Ergonomics
Brief Title: Safety Voice for Ergonomics as a Preventive Approach for Work-related Musculoskeletal Disorders in Masonry Apprentices
Acronym: SAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eastern Washington University (Other)
Collaborators: Oregon State University (Other); University of Oregon (Other); St. Luke's Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Daniel Anton, Principal Investigator, Eastern Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2U60OH009762-06 (NIH)
Record Dates: First submitted 2016-01-28; First posted 2016-02-08 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Work Related Musculoskeletal Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ergonomics Training Only (Experimental): Participants in this arm receive Ergonomics training only
  Interventions: Behavioral: Ergonomics training and/or Safety Voice training
- Ergonomics and Safety Voice Training (Experimental): Participants in this arm receive training on both Ergonomic principles and Safety Voice training
  Interventions: Behavioral: Ergonomics training and/or Safety Voice training
- Control Group (No Intervention): Participants in this arm will receive no additional Ergonomics or Safety Voice training

INTERVENTIONS:
Behavioral: Ergonomics training and/or Safety Voice training — Ergonomics training will focus on ergonomic principles specific to masonry such as goals of ergonomics, common musculoskeletal disorders among masons, modifiable work factors and risk factors, hazard analysis, hierarchy of controls, and current ergonomic solutions for masonry. Safety Voice training will focus on development of skills such as self-direction, self-control, accountability, responsibility, communication strategies, and leadership that can help them to develop a "safety voice" about safety in general, and ergonomics specifically.
  Arms: Ergonomics Training Only; Ergonomics and Safety Voice Training

SUMMARY:
Masons have the highest rate of overexertion injuries among all construction trades and rank second as an occupation for back injuries in the United States. Identified ergonomic solutions are the primary method of reducing exposure to risk factors associated with musculoskeletal disorders. However, many construction workers lack knowledge about these solutions, as well as basic ergonomic principles. Construction apprentices, as they embark on their careers, are greatly in need of ergonomics training to minimize the cumulative exposure that leads to musculoskeletal disorders. Apprentices receive safety training; however, ergonomics training is often limited or non-existent. In addition, apprenticeship programs often lack "soft skills" training on how to appropriately respond to work environments and practices that are unsafe. The SAVE program - SAfety Voice for Ergonomics - strives to integrate evidence-based health and safety training strategies into the mason apprenticeship skills training to teach ergonomics, problem solving, and speaking up to communicate solutions that reduce musculoskeletal injury risk. The central hypothesis is that the combination of ergonomics training and safety voice promotion will be more effective than no training or either ergonomics training alone or safety voice training alone.

Following the development and pilot testing of the SAVE intervention, SAVE will be evaluated in a cluster-randomized controlled trial at 12-15 masonry training centers across the U.S. Clusters of apprentices within centers will be assigned at random to one of three intervention groups (n = 32 per group): (1) ergonomics training only, (2) combined ergonomics and safety voice training, or (3) control group with no additional training intervention. Outcomes assessed at baseline, at the conclusion of training, and then at six and 12 months post training will include: musculoskeletal symptoms, general health perceptions, knowledge of ergonomic and safety voice principles, and perception and attitudes about ergonomic and safety voice issues.

DETAILED DESCRIPTION:
A. Rationale Masons have the highest rate of overexertion injuries among all construction trades and rank second as an occupation for back injuries in the United States. Identified ergonomic solutions are the primary method of reducing exposure to risk factors associated with musculoskeletal disorders. However, many construction workers lack knowledge about these solutions, as well as basic ergonomic principles. Construction apprentices have the greatest need for ergonomics training as they embark on their careers to minimize cumulative exposure that leads to musculoskeletal disorders. Additionally, apprenticeship training programs often lack "soft skills" training on how to appropriately respond to work environments and practices that are unsafe. The SAVE program - SAfety Voice for Ergonomics - strives to integrate evidence-based health and safety training strategies into current masonry apprenticeship skills training to teach ergonomics, problem solving, and speaking up to reduce musculoskeletal injury risk. SAVE will incorporate blended learning principles by combining traditional, face-to-face teaching methods with e-learning methods.

B. Objectives The primary objective of this project is to evaluate the SAVE program in a cluster randomized controlled trial in 12-15 masonry training centers. Clusters of apprentices within centers will be assigned at random to one of four intervention groups (n = 32 per group): (1) ergonomics training only, (2) combined ergonomics and safety voice training, or (3) control group with no additional training intervention. Outcomes assessed at baseline, at the conclusion of training, and then at 6 and 12 months post training will include: musculoskeletal symptoms, general health perceptions, knowledge of ergonomic and safety voice principles, and perception and attitudes about ergonomic and safety voice issues. The central hypothesis is that the combination of ergonomics training and safety voice promotion will be more effective than no training or either ergonomics training alone or safety voice training alone.

C. Procedures Primary Training Program E-learning Modules. Depending on the group to which a training center is assigned, apprentices within that center will view brief e-learning training modules to provide apprentices with basic knowledge of ergonomic and/or safety voice principles. These modules include text, brief video clips, and interactive on-screen slides that guide apprentices through content with brief quizzes that assure understanding. Apprentices will complete the modules at the apprenticeship training center. Learning gained from completing the e-learning modules will be reinforced by short (10-20 minute), applied, face-to-face experiential activities. These interactive, face-to-face, problem-solving activities will complement the e-learning and will include vignettes to promote discussion of hypothetical worksite cases related to ergonomics and/or safety voice. These vignettes will be brief to fit into existing training time demands.

Secondary (Refresher) Training Program Refresher training for ergonomics and/or safety voice will bolster concepts learned by apprentices in the primary training. Depending on the group to which a training center is assigned, apprentices within that center will receive refresher training through text messages that are sent by the researchers. Secondary training is considered medium engagement learning since apprentices will respond to texts. For example, an ergonomic-related text message would read, "Keeping work between knee and shoulder level reduces the risk of a back or shoulder injury. During the past week have you worked on adjustable scaffolding?" The apprentice will respond "Yes" or "No." Apprentices responding "Yes" will receive a follow-up text/email reminding them of the importance of keeping work between knee and shoulder level. Refresher training will be delivered over a one-year period to maximize knowledge retention.

ELIGIBILITY:
Inclusion Criteria:

* Currently employed masonry apprentices in their first two years of training and at least 18 years of age will be recruited to participate and provide signed informed consent. No potential participant will be excluded because of co-morbid medical conditions.

Exclusion Criteria:

* Apprentices who do not have reliable access to a computer or who do not use a cell phone will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Modified Nordic Questionnaire | Change from baseline through study completion, an average of 1 year
  The Modified Nordic Questionnaire assesses self-reported musculoskeletal symptoms. The questionnaire requires a "yes" or "no" response to three questions for nine different anatomic sites: "During the last 12 months have you had a job-related ache, pain, discomfort"; "During the last 12 months have you been prevented from doing your day's work due to this condition?" and "During the last 12 months have you seen a physician for this condition?"
Short Form-36 Health Survey (SF-36v2®) | Change from baseline through study completion, an average of 1 year
  The Short Form-36 Health Survey (SF-36v2®) is a standardized health questionnaire of perceived physical and mental health status, which has been shown to be associated with occupational safety and health behavior change.
SAVE Reaction | Change from baseline through study completion, an average of 1 year
  To measure the reaction of the apprentices to the SAVE training, four, standard, 5-point scale questions will be used (1 = strongly disagree to 5 =strongly agree).
SAVE Knowledge Acquisition | Change from baseline through study completion, an average of 1 year
  These questions will assess knowledge gained of ergonomic and safety voice principles covered in the SAVE program.
SAVE Attitude, Compliance, and Participation | Change from baseline through study completion, an average of 1 year
  These questions will evaluate apprentice attitudes and perception about ergonomic and safety voice issues using a 5-point scale (strongly disagree to strongly agree).
SAVE Adoption | Change from baseline through study completion, an average of 1 year
  These questions will provide information about whether apprentices used interventions more frequently, or were more willing to adopt new ergonomic interventions when appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Washington University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kincl LD, Anton D, Hess JA, Weeks DL. Safety voice for ergonomics (SAVE) project: protocol for a workplace cluster-randomized controlled trial to reduce musculoskeletal disorders in masonry apprentices. BMC Public Health. 2016 Apr 27;16:362. doi: 10.1186/s12889-016-2989-x. PMID 27121123